CLINICAL TRIAL: NCT00871390
Title: Complex Electrograms in Atrial Fibrillation: Spatiotemporal Organization and Mechanistic Insights and Organization in Acute Atrial Fibrillation Post Open Heart Surgery
Brief Title: Organization of Excitation in People With Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Omer Berenfeld, Associate Professor of Internal Medicine and Biomedical Engineering, University of Michigan
Other Study IDs: 628; P01HL039707 (NIH)
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Atrial Fibrillation
Keywords: Paroxysmal Atrial Fibrillation; Permanent/Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Biopsys
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Atrial fibrillation (AF) is a condition in which the upper chambers of the heart, the atria, undergo an irregular beating rhythm. Despite the fact that AF is the most common type of sustained cardiac rhythm disturbance the investigators still do not understand it entirely and its current therapies are only marginally effective. The overall goal of our project is to determine the organization and mechanisms of electrical activation patterns during AF in humans.

DETAILED DESCRIPTION:
Experiments in animal hearts demonstrated that some cases of atrial fibrillation (AF) may be maintained by a small number of drivers in the form of self-sustained, reentrant, electrical impulses located in the posterior left atrium (LA) wall, near the pulmonary veins (PV/LA junction). In those experiments, the fastest rotors acted as the highest frequency drivers that maintained the overall activity. This resulted in a hierarchy of local excitation frequencies throughout both atria. More recently, clinical studies have confirmed the existence of a hierarchical organization in the rate of activation of different regions in the atria of patients with paroxysmal and chronic atrial fibrillation. However, the mechanisms underlying such a hierarchical distribution of frequencies in human AF has not been explored. Our project will try to demonstrate the general hypothesis that both local activation frequency and degree of regularity, while different in different parts of the atrium, are distributed non-randomly, with different patterns of distribution in paroxysmal versus chronic AF patients. We further surmise that such patterns are the result of interrupted propagation of impulses emanating from the drivers localized at the site of highest frequency and organization activity, with a gradual reduction of activation frequency as the distance from the driver increases. To test our hypotheses we will use a combination of clinical and numerical studies. For the clinical part we will gather patients data in a collaborative site at Rochester, NY. The data obtained in that site will be analyzed and interpreted at the Institute for Cardiovascular Research in SUNY Upstate Medical University. For the numerical part, simulations on computer models of AF will be performed solely in the Institute for Cardiovascular Research. Our Specific Aims are: 1. Characterize the frequency of activation during AF in patients after heart surgery and relate it to the presence of fibrosis. 2. In computer simulations, to study the mechanisms of initiation and maintenance of AF at the PV/LA junction using three different computer models with increasing anatomical complexity (the description of the computer simulations is available only in the grant application). Successful achievement of our specific aims should help us advance understanding of the mechanisms and manifestations of this complex arrhythmia and may help to directly improve the efficacy of pharmacological and ablative therapies of AF in patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical indication for curative ablation of AF
* Patients will be enrolled as they are referred for the ablation therapy or post open heart surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with paroxysmal and chronic atrial fibrilation (AF).
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2006-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Omer Berenfeld, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - SUNY Upstate Medical University, Syracuse, New York